CLINICAL TRIAL: NCT04534712
Title: Lymphocyte - Monocyte Ratio As An Independent Predictor For Progression Of Illness In Patients With Covid-19
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, VAMSIDHAR, DNB Trainee, Sir Ganga Ram Hospital
Other Study IDs: yet to be assigned
Record Dates: First submitted 2020-08-30; First posted 2020-09-01 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Covid19
Keywords: LYMPHOCYTE MONOCYTE RATIO; COVID-19; DISEASE PROGRESSION
MeSH Terms: conditions — COVID-19; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PROGRESSION: Cohort A with patients who progressed to next stage of illness or continue to remain in the same stage
  Interventions: Diagnostic Test: LYMPHOCYTE MONOCYTE RATIO
- NON PROGRESSION: Cohort B with those who improved by two points on the ordinal scale without any further progression
  Interventions: Diagnostic Test: LYMPHOCYTE MONOCYTE RATIO

INTERVENTIONS:
Diagnostic Test: LYMPHOCYTE MONOCYTE RATIO — Absolute lymphicyte and absolute monocyte counts are recorded on admission of COVID -19 positive patient and ratio is derived. the patients are followed up for any progression of disease stage.

SUMMARY:
Corona virus disease 2019 (COVID 19), first identified in December 2019 in a cluster of population in a Chinese province, soon emerged as a pandemic, causing a huge strain on healthcare system and mortality all over the world. An ideal marker for predicting course of this illness should be easily available and reproducible; as the disease burden has spread to third world countries whose healthcare system is resource limited. Our study is aimed to study the utility of lymphocyte- monocyte ratio in the early stages to predict the progression of COVID 19 pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* All adults of age 18-80 years tested positive for SARS-CoV-2 reverse-transcriptase - polymerase chain reaction (rt-PCR) and presented within 7 days of symptom(s) onset

Exclusion Criteria:

* Pregnancy
* Sepsis
* Malignancy
* Patients on immunosuppressant therapy
* Chronic inflammatory conditions
* Cases lost to follow up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who are tested positive for COVID 19 and presented within 7 days of symptom onset will be included
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
progression | 28 days
  disease progression equal or more than 2 stages

SECONDARY OUTCOMES:
mortality | 28 days
  end outcome of the patients diagnosed of COVID-19 infection

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
IPD data shall be shared on request basis.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 1 year from the study completion till publication